CLINICAL TRIAL: NCT07232017
Title: Implementation of Intensive Hypertension Management Approaches: Cleveland Clinic
Acronym: IN-HOME BP
Status: Recruiting | Type: Observational
Sponsor: Anita Misra-Hebert (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Anita Misra-Hebert, Professor of Medicine, Cleveland Clinic Lerner College of Medicine of Case Western Reserve University, Staff, Department of Internal Medicine, Director, Healthcare Delivery and Implementation Science Center, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 25-792
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hypertension (HTN)
Keywords: hypertension; uncontrolled blood pressure; home blood pressure; pharmacist; advanced practice provider
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IN-HOME BP: titrating BP medications based on patient-recorded home blood pressure readings: This project will utilize evidence from a randomized controlled trial by Margolis et al.(1) to build upon Cleveland Clinic's existing team-based primary care provider (PCP) collaboration with pharmacists and advanced practice providers (APP) and will use a mechanism that allows titrating blood pressure medications based on patient-recorded home blood pressure readings.
  Interventions: Other: IN-HOME BP

INTERVENTIONS:
Other: IN-HOME BP — A team-based approach with a primary care provider (PCP) collaborating with pharmacists and advanced practice providers (APP) and will use a mechanism (frequent follow-up- phone or virtual appointments) that allows titrating blood pressure medications based on patient-recorded home blood pressure readings.

SUMMARY:
The primary objective of the Implementation of Effective Hypertension Management Approaches: Cleveland Clinic program is to improve blood pressure control for patients diagnosed with hypertension (HTN) and uncontrolled blood pressure, specifically defined as a blood pressure greater than 150/95, across all Cleveland Clinic Northeast Ohio primary care practices. The project will scale up the availability of resources for treating hypertension in 56 primary care practices within the Cleveland Clinic Health System in Northern Ohio, reaching up to approximately 3800 patients. This project will utilize evidence from a randomized controlled trial by Margolis et al.(1) to build upon Cleveland Clinic's existing team-based primary care provider (PCP) collaboration with pharmacists and advanced practice providers (APP) and will use a mechanism that allows titrating blood pressure medications based on patient-recorded home blood pressure readings.

DETAILED DESCRIPTION:
Primary care providers will offer the program to patients in Northeast Ohio with a hypertension diagnosis and aged 18-85, except those who are pregnant, have stage 5 chronic kidney disease or end stage renal disease, or enrolled in hospice care. The project time frame is 48 months. Quantitative and qualitative methods will be used to evaluate implementation and effectiveness outcomes associated with the program. Electronic medical records and surveys will be the key data sources for the quantitative evaluation. Qualitative data collection methods will include semi-structured interviews, field observations, and periodic reflections.

Specific Aims Aim 1. To prepare for implementation of the intensive HTN management program across all Northeast Ohio Primary Care Practices (Pre-Implementation) Pre-Implementation Phase (12 months)

* Quantitative assessment of practice variation in HTN control.
* Qualitative assessment of practice barriers and facilitators to HTN management.
* Creation of a clinical decision support tool for program referral.
* Creation of project-specific patient and employee Advisory Panel.
* Pharmacist and advanced practice provider (APP) training for delivery of the program.
* Practice facilitation training with the Cleveland Clinic continuous improvement team.
* Community Health Worker/Primary Care Navigator Training for Patient Outreach.
* Creation of presentations for primary care staff meetings. Aim 2. To implement the intensive HTN management program across all Northeast Ohio Primary Care Practices (Rollout and Active Implementation) Implementation Phase (24 months)
* Stepped wedge rollout of intensive HTN management program.
* Implementation of the clinical decision support tool at implementation sites.
* Community Health Worker/Primary Care Navigator outreach to patients.
* Delivery of Presentations at primary care staff meetings.
* Practice Facilitation at Implementation Sites.
* Qualitative data collection regarding patient and provider implementation outcomes of acceptability and feasibility.
* Quantitative data collection of implementation outcomes of adoption, fidelity, effectiveness, implementation cost; provider surveys re: acceptability, appropriateness, feasibility.
* Patient and employee advisory panel input into implementation evaluation. Aim 3. To monitor and evaluate the maintenance of the intensive HTN management program across all Northeast Ohio Primary Care Practices (Maintenance) Maintenance Phase (9 months)
* Quantitative data collection of implementation outcomes-reach, adoption, fidelity, effectiveness, cost-compared to the active implementation phase.
* Capture practice-level adaptations with comparison to the active implementation phase.
* Complete final data collection and analyses.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis, aged 18-85 years old
* Uncontrolled blood pressure, defined as a blood pressure reading of > 150/95

Exclusion Criteria:

* pregnant, stage 5 chronic kidney disease, End Stage Renal Disease, enrolled in hospice care

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Per inclusion criteria and that the patient has at least 2 encounters with a HTN diagnosis within the past 24 months; had an encounter within the past 12 months at their PCPs assigned location; had a documented systolic blood pressure of >150 or diastolic blood pressure of >95 at the most recent encounter at the primary care location, and a previous encounter within the health system within the past 24-month qualifying time frame with a documented systolic blood pressure of >150 or diastolic blood pressure of >95.
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure Change | Patients will be followed for up to 33 months: 24-month implementation/intervention period and 9-month maintenance period.
  The main effectiveness finding the investigators expect to report at the end of the proposed implementation project is the change in patient systolic blood pressure from baseline to 12 months post-implementation. The expected change in systolic blood pressure based upon Margolis et al.(1) is -18mmHg. The period of evaluation will be from the time of program enrollment, with home BP measurements assessed every 2-3 weeks until the blood pressure is less than 135/85 and at 12 months. The blood pressure will continue to be measured every 6 months through the full the 24-month implementation/intervention period (allowing all sites to roll out the intervention) and a 9-month maintenance period.

SECONDARY OUTCOMES:
Diastolic Blood Pressure Change | The patient's blood pressure will be measured for up to 33 months (24-month implementation/intervention period and 9-month maintenance period). Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance.
  Change in the patient's diastolic blood pressure from baseline as measured in mmHg.
Reach (Actual): Patients Offered, Initiated, Completed | Measured every 3 months for up to 33 months.
  Number of patients who were offered, who initiated, and completed the intensive HTN intervention program. Measured by total number at sorted by each: offered, initiated, completed.
Effectiveness: Equity in Outcomes (Race) | Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance: for up to 33 months.
  Blood pressure change stratified by demographic factors, specifically race. Measured as percentage of black, white, and other.
Effectiveness: Equity in Outcomes (Ethnicity) | Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance: for up to 33 months.
  Blood pressure change stratified by demographic factors, specifically ethnicity. Measured by percentage of Hispanic and non-Hispanic
Effectiveness: Equity in Outcomes (Gender) | Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance: for up to 33 months.
  Blood pressure change stratified by demographic factors, specifically gender. Measured by percentage of male and female.
Effectiveness: Equity in Outcomes (Age) | Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance: for up to 33 months.
  Blood pressure change stratified by demographic factors, specifically age group. Measured in years.
Effectiveness: Equity in Outcomes (Insurance) | Every 2-3 weeks during intervention, at 12 months, then every 6 months through maintenance: for up to 33 months.
  Blood pressure change stratified by demographic factors, specifically insurance. Measured in number of insurance: Medicare, Medicaid, Commercial, Self-pay.
Effectiveness: Medication change | Every 2-3 weeks during intervention then every 6 months through maintenance: for up to 33 months.
  Change from baseline medication regimen (medication class and dosage).
Effectiveness: Medication Adherence | Every 2-3 weeks during intervention then every 6 months through maintenance: for up to 33 months.
  Pharmacy Fill Data
Effectiveness: Cardiovascular outcomes | Baseline, and every 6 months through maintenance: for up to 33 months.
  Sustained blood pressure control resulting in decreased cardiovascular risk: reported myocardial infarction, acute coronary syndrome, stroke, heart failure, arrhythmia, and death.
Effectiveness: Acute Renal Failure - Change in glomerular filtration rate (GFR). | Every 6 months through maintenance: for up to 33 months.
  Assessing acute renal failure by change in glomerular filtration rate (GFR) as measured in milliliters/minute/1.73 meters squared.
Effectiveness: PROMIS-10 Survey | Baseline at intake visit then at 12 months: up to 24-months.
  See improvement of patient report outcomes captured at pre-visit PROMIS-10 survey(12) administration as part of routine clinical care. As measured by assessing scores over time.
Effectiveness: Adverse Effects | Every 2-3 weeks during intervention then every 6 months through maintenance: for up to 33 months.
  Patient reported adverse effects at follow-up visits during intervention. Measured as number of effects reported by patient.
Implementation: Provider views of the Acceptability, Appropriateness, and Feasibility survey | Every 6 months starting throughout active implementation and maintenance: for up to 33 months.
  Captured through surveys, provider views of Acceptability, Appropriateness, Feasibility (13). Providers views of intervention may impact adoption of intervention for patients. Measured by change in item scored over time.
Primary Care Provider Adoption | Every 3 months during intervention period: for up to 24 months
  Number of providers in each practice group referring to the Intensive HTN program will be measured by the number of referrals attributed to practice group.
Pharmacist Adoption | Every 3 months during intervention period: for up to 24 months.
  Number of patients in the program attributed to the trained pharmacy providers eligible to deliver the program.
Advanced Practice Provider Adoption | Every 3 months during intervention period: for up to 24 months.
  Number of patients in the program attributed to the trained Advanced Practice Providers (APP) eligible to deliver the program.
Formal Qualitative Assessment of context of high proportion of HTN control and low proportion of HTN control practices: Pre-Implementation | Pre-Implementation: up to 12 months.
  To understand barriers and facilitators to achieving HTN control
  * Semi-structured interviews with non-patient (employee) key stakeholders at practices with high/low proportion of HTN control
  * Direct field observations of high-low referral practice sites Qualitative methodologists will analyze the qualitative data (transcripts and descriptive fieldnotes) will be coded to reflect key domains of interest and emergent themes.
Formal Qualitative Assessment: Observations of Employee and Patient Advisory Panels | Quarterly meetings throughout pre- and active implementation: up to 36 months.
  To examine anticipated barriers and facilitators to implementation and to assess ongoing implementation activities. Qualitative methodologists will analyze the qualitative data (fieldnotes) will be coded to reflect key domains of interest and emergent themes.
Formal Qualitative Assessment: Semi-structured Interviews with Patients at High/Low proportion of HTN Control | Baseline, 6 months, 12 months during active implementation: up to 24 months.
  Inviting a sample of patients receiving the intervention at high and low proportion of HTN control practices to participate in interviews to assess perceptions of acceptability of the intensive HTN management program.
  Qualitative methodologists will analyze the qualitative data (transcripts) will be coded to reflect key domains of interest and emergent themes.
Formal Qualitative Assessment: Periodic Reflections with agents of implementation | Monthly or bimonthly throughout active implementation and maintenance: for up to 33 months.
  Periodic reflections conducted with a subgroup of pool of primary care providers, pharmacists, and APPs across practice locations to understand barriers and facilitators to achieving hypertension control.
  Qualitative methodologists will analyze the qualitative data (descriptive fieldnotes) will be coded to reflect key domains of interest and emergent themes.
Outcome measure type: Effectiveness (Hospitalizations / Emergency Department Visits) | Every 6 months: up to 33 months.
  Hospitalizations and Emergency Department Visits: number of acute care hospitalizations, number of emergency department visits. Determining association between intensive HTN management and acute care utilization.
Outcome Measure Type: Effectiveness (Outpatient Visits) | Every 6 months: up to 33 months.
  Outpatient visits other than for the intensive HTN management program. Number of outpatient visits (in-clinic or virtual, primary care and specialty). To determine association between intensive HTN management and acute care utilization.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data used for this study includes human research participant data that are sensitive and cannot be publicly shared due to legal and ethical restrictions by the Cleveland Clinic regulatory bodies, including the institutional review board and legal counsel. We will make our data sets available on request, under appropriate data use agreements with the specific parties interested in academic collaboration.

REFERENCES:
- [Background] Cuttaree P, Edlund G, Eriksson M, Granberg P, Lager O, Lonberg E, Sjoberg P, Widell K. [Should sick children be kept in bed?]. Lakartidningen. 1971 Mar 24;68(13):1485-8. No abstract available. Swedish. PMID 5576104
- [Background] Murakami K, Minoshima S, Uno K, Arimizu N, Kobayashi M, Fujita M, Okamoto S, Ikehira H, Fukuda H, Tateno Y. [Imaging of malignant melanoma with In-111-labeled monoclonal antibody (ZME-018) and Ga-67 scintigraphy]. Kaku Igaku. 1989 Jan;26(1):113-9. No abstract available. Japanese. PMID 2724630
- [Background] Margolis KL, Bergdall AR, Crain AL, JaKa MM, Anderson JP, Solberg LI, Sperl-Hillen J, Beran M, Green BB, Haugen P, Norton CK, Kodet AJ, Sharma R, Appana D, Trower NK, Pawloski PA, Rehrauer DJ, Simmons ML, McKinney ZJ, Kottke TE, Ziegenfuss JY, Williams RA, O'Connor PJ. Comparing Pharmacist-Led Telehealth Care and Clinic-Based Care for Uncontrolled High Blood Pressure: The Hyperlink 3 Pragmatic Cluster-Randomized Trial. Hypertension. 2022 Dec;79(12):2708-2720. doi: 10.1161/HYPERTENSIONAHA.122.19816. Epub 2022 Oct 25. PMID 36281763